CLINICAL TRIAL: NCT00265109
Title: Open-Label Study of Levetiracetam in Body Dysmorphic Disorder
Brief Title: Effectiveness of Levetiracetam in the Treatment of Body Dysmorphic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0410-001
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Body Dysmorphic Disorder
Keywords: body dysmorphic disorder; levetiracetam
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Levetiracetam

ARMS (1):
- open label (Other): Open-label trial; all participants received levetiracetam
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — The initial levetiracetam dose will be 250 mg/day, which will be increased to 250 mg BID after 1 week. The dose will then be increased by 500 mg/day each week (given in BID dosing) to a maximum of 3,000 mg/day. The dose will be raised more slowly or the maximum dose will not be reached if response occurs at a lower dose or side effects are problematic. Subjects who are unable to tolerate at least 500 mg a day of levetiracetam will be withdrawn from the study.

SUMMARY:
The purpose of this study is to assess the usefulness of a medication (Levetiracetam) for people with body dysmorphic disorder.

DETAILED DESCRIPTION:
Body dysmorphic disorder (BDD), a perceived defect in appearance (e.g., a "large" nose or facial "scarring"), is a relatively common disorder that causes marked distress and impairment in functioning. Recent data suggests that adults with BDD may respond to serotonin reuptake inhibitors (SRIs); however, response to SRIs is often only partial. About one third of patients do not respond to an SRI. Furthermore, patients may stop taking SRIs because of side effects (e.g., sexual side effects). For these reasons, additional monotherapy and SRI augmentation strategies are greatly needed.

Levetiracetam is primarily used as an antiseizure medication and has a wider safety margin than other antiepileptics. Preliminary scientific studies may suggest that it may be helpful for certain psychiatric symptoms and disorders. In the present study we propose to obtain pilot data on 1) levetiracetam monotherapy and 2) levetiracetam augmentation of SRIs in patients with BDD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65;
* Current DSM-IV BDD or its delusional variant (delusional disorder, somatic type) for at least 3 months;
* A minimum total score of 20 on the Yale-Brown Obsessive Compulsive Scale Modified for BDD (BDD-YBOCS) (19);
* Suitable for treatment in an outpatient setting

Exclusion Criteria:

* Unstable medical illness, including renal failure or dialysis;
* Myocardial infarction within 6 months;
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
* A need for prn benzodiazepines, another antiepileptic medication, or an anticipated change in the dose of any concomitant medications while receiving treatment with levetiracetam;
* Clinically significant suicidality, including a suicide attempt within the past two months;
* Lifetime history of DSM-IV dementia, schizophrenia, or any other DSM-IV psychotic disorder that is not attributable to BDD;
* Current or recent (past 3 months) DSM-IV substance abuse or dependence;
* Initiation of ongoing psychotherapy from a mental health professional within 3 months prior to study baseline;
* Ongoing cognitive-behavioral therapy from a mental health professional;
* Previous treatment with levetiracetam;
* Treatment with investigational medication, depot neuroleptics, or ECT within the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A Phillips, M.D., Principal Investigator — Rhode Island Hospital/ Brown University
Locations (1):
- Rhode Island Hospital Body Dysmorphic Disorder Program, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study — http://www.bodyimageprogram.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Levetiracetam: All 17 participants in the study received Levetiracetam. The initial dose was 250 mg/day, which was increased to 250 mg BID after 1 week. The dose was then increased by 500 mg/day each week (given in BID dosing) to a maximum of 3,000 mg/day. The dose was raised more slowly or the maximum dose was not reached if response occurred at a lower dose or side effects were problematic.
Period: Overall Study
Arm/Group | Open-Label Levetiracetam
Started | 17
Completed | 11
Not Completed | 6
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders on the Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS)
Description: The BDD-YBOCS, a reliable and valid 12-item semi-structured clinician-administered scale assessed BDD severity during the past week. 38 items are rated from 0 (no symptoms) to 4 (extreme symptoms); range=0-48. This scale assesses preoccupation with the perceived appearance defects, associated compulsive behaviors, insight, and avoidance. A ≥30% decrease in total score indicated response.
Time Frame: Baseline to end week 12
Population: Analyses of the primary outcome measure were intention to treat (ITT) analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
Participants | 9

2. Secondary Outcome: Percentage of Participants Who Improved on the Body Dysmorphic Disorder Clinical Global Impressions Scale - Clinician Rating for BDD Symptoms
Description: The Clinical Global Improvement Scale (CGI) is a widely used 7-point scale that assesses global improvement or worsening of symptoms, with ratings ranging from "very much worse" (score of 7) to "very much improved" (score 1). Ratings of much improved (score of 2) or very much improved (score of 1) defined improvement in BDD.
Time Frame: Last week of treatment (week 12) or last week of treatment for early dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 17
Participants | 8

3. Secondary Outcome: Percentage of Subjects Who Improved on the Clinical Global Improvement Scale (CGI) -- Clinician Rating of Global Improvement.
Description: The CGI is a widely used 7-point scale that assesses global improvement or worsening of symptoms, with ratings ranging from "very much worse" (score of 7) to "very much improved" (score 1). Ratings of much improved (score of 2) or very much improved (score of 1) defined global improvement.
Time Frame: Last week of treatment (week 12)
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 17
Participants | 9

4. Secondary Outcome: Percentage of Participants Who Improved on the Body Dysmorphic Disorder Clinical Global Impressions Scale - Patient Rating for BDD Symptoms
Description: as for outcome 2
Time Frame: Last week of treatment (week 12) or last week of treatment for early dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 17
Participants | 8

5. Secondary Outcome: Percentage of Subjects Who Improved on the Clinical Global Improvement Scale (CGI) -- Patient Rating of Global Improvement.
Description: as for outcome 3
Time Frame: Last week of treatment (week 12)
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 17
Participants | 8

6. Secondary Outcome: Scores on Brown Assessment of Beliefs Scale
Description: The Brown Assessment of Beliefs Scale (BABS) is a 7-item semi-structured clinician-administered scale that assesses seven components of delusionality (insight) during the past week. Scores range from 0-24, with higher scores indicating greater delusionality. Beliefs are also categorized as delusional or nondelusional using an empirically derived cutpoint.
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 14.6 (4.3)
  Post-treatment | 10.4 (5.3)

7. Secondary Outcome: Scores on Clinical Global Severity
Description: The 7-point Clinical Global Severity Scale assessed current illness severity at study baseline (score of 1=normal, not at all ill, and score of 7=among the most extremely ill patients).
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 5.2 (1.0)
  Post-treatment | 4.2 (1.6)

8. Secondary Outcome: Scores on Hamilton Depression Rating Scale
Description: The 24-item Hamilton Rating Scale for Depression (HAM-D 24) is a widely used reliable and valid clinician-administered measure of current severity of depressive symptoms. Scores range from 0 to 76, with higher scores reflecting more severe depressive symptoms.
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 18.1 (6.4)
  Post-treatment | 11.4 (8.4)

9. Secondary Outcome: Scores on Beck Anxiety Inventory
Description: The Beck Anxiety Inventory (BAI) is a reliable, valid, and widely used 21-item self-report measure of anxiety during the past week which focuses on somatic symptoms.44 The BAI has been shown to be sensitive to change. Scores range from 0-63, with higher scores reflecting more severe symptoms.
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 12.4 (6.8)
  Post-treatment | 9.6 (5.5)

10. Secondary Outcome: Scores on Social Phobia Inventory
Description: The Social Phobia Inventory (SPIN) is a 17-item self-report questionnaire that assesses fear, avoidance, and physiological arousal associated with social anxiety during the past week. This scale is reliable, valid, and sensitive to change. Scores range from 0-68, with a score ≥19 distinguishing patients with social phobia from both healthy controls and psychiatric controls without social phobia.
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 32.9 (12.4)
  Post-treatment | 29.4 (13.8)

11. Secondary Outcome: Scores on Global Assessment of Functioning
Description: The Global Assessment of Functioning (GAF) is a global measure of symptom severity and psychological, social, and occupational functioning. Scores range from 0-100, with lower scores denoting more severe illness and/or poorer functioning
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 46.1 (7.8)
  Post-treatment | 55.8 (14.5)

12. Secondary Outcome: Scores on Social and Occupational Functioning Scale (SOFAS)
Description: The Social and Occupational Functioning Scale (SOFAS) is a global measure of psychological, social, and occupational functioning. Scores range from 0-100, with lower scores denoting more severe illness and/or poorer functioning
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 47.0 (8.5)
  Post-treatment | 59.8 (18.6)

13. Secondary Outcome: Scores on The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) -- Short Form
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q), Short Form, is a 14-item reliable and valid measure that is sensitive to change. Transformed scores range from 0 from 100, with lower scores reflecting poorer quality of life.The Short Form transformed score is reported.
Time Frame: Pre- and post-treatment (week 12)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Levetiracetam
Number analyzed (Participants) | 17
units on a scale
  Pre-treatment | 49.5 (10.3)
  Post-treatment | 57.4 (14.8)

ADVERSE EVENTS:
Arm/Group | Open-Label Levetiracetam
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Levetiracetam (N=17)
Increased depression and suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Levetiracetam (N=17)
Fatigue (Psychiatric disorders) | 8 (8)
Irritability (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4)
Headache (Psychiatric disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Nausea (Psychiatric disorders) | 2 (2)
Dizziness (Psychiatric disorders) | 2 (2)
Feelings of Detachment (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Back Aches (Psychiatric disorders) | 1 (1)
Constipation (Psychiatric disorders) | 1 (1)
Decreased Libido (Psychiatric disorders) | 1 (1)
Diarrhea (Psychiatric disorders) | 1 (1)
Dyspepsia (Psychiatric disorders) | 1 (1)
Forgetfulness (Psychiatric disorders) | 1 (1)
Muscle Aches (Psychiatric disorders) | 1 (1)
Feeling Depressed (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a small open-label trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No